CLINICAL TRIAL: NCT03426449
Title: Posterolateral Versus Lateral Internal Anal Sphincterotomy for Chronic Anal Fissure: A Randomized Clinical Trial
Brief Title: Posterolateral Versus Lateral Internal Anal Sphincterotomy for Chronic Anal Fissure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Sameh Emile, Lecturer of general surgery, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: mansourau45
Record Dates: First submitted 2018-02-02; First posted 2018-02-08 (Actual); Last update posted 2018-02-09 (Actual); Status verified 2018-02

CONDITIONS: Anal Fissure
MeSH Terms: conditions — Fissure in Ano | interventions — Lateral Internal Sphincterotomy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Posterolateral sphincterotomy (Active Comparator): Division of internal anal sphincter at 5 o'clock position
  Interventions: Procedure: posterolateral sphincterotomy
- Lateral sphincterotomy (Active Comparator): Division of internal anal sphincter at 3 o'clock position
  Interventions: Procedure: lateral sphincterotomy

INTERVENTIONS:
Procedure: posterolateral sphincterotomy — Fissurectomy and limited division of internal anal sphincter at 5 o'clock position for 8-10 mm
  Arms: Posterolateral sphincterotomy
Procedure: lateral sphincterotomy — Fissurectomy and limited division of internal anal sphincter at 3 o'clock position for 8-10 mm
  Arms: Lateral sphincterotomy

SUMMARY:
The present study aimed to compare the standard lateral internal sphincterotomy at 3 o'clock with posterolateral internal sphincterotomy at 5 o'clock in regards healing time, postoperative recurrence and complications, particularly fecal incontinence.

DETAILED DESCRIPTION:
The present study aimed to compare the standard lateral internal sphincterotomy at 3 o'clock with posterolateral internal sphincterotomy at 5 o'clock in regards healing time, postoperative recurrence and complications, particularly fecal incontinence. We hypothesized that performing internal sphincterotomy in a point midway between the standard lateral position and the posterior midline position would confer better healing and relief of symptoms with less incidence of fecal incontinence while avoiding the development of keyhole deformity.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of both genders with chronic posterior anal fissure were included to the study.

Exclusion Criteria:

* Patients with anterior or lateral anal fissure,
* patients with previous anal surgery,
* patients with concomitant anorectal pathology,
* patients with secondary anal fissure due to Crohn's disease or other specific etiology,
* patients with any degree of fecal incontinence,
* patients with active anorectal sepsis.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-07-30 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Duration of healing | 6-8 weeks after surgery
  The time to complete healing of anal wound defined by complete epithelization of the wound

SECONDARY OUTCOMES:
Anal pain | 1-6 weeks after surgery
  Degree of postoperative pain assessed by pain visual analogue scale ranging from 0-10 where 0 indicates no pain and 10 indicates the worst possible pain

CONTACTS AND LOCATIONS:
Overall Officials: Sameh H Emile, M.D., Principal Investigator — Mansoura University Hospital
Locations (1):
- Mansoura university hospital, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alawady M, Emile SH, Abdelnaby M, Elbanna H, Farid M. Posterolateral versus lateral internal anal sphincterotomy in the treatment of chronic anal fissure: a randomized controlled trial. Int J Colorectal Dis. 2018 Oct;33(10):1461-1467. doi: 10.1007/s00384-018-3087-6. Epub 2018 May 19. PMID 29779044